CLINICAL TRIAL: NCT06276322
Title: Assessment and Comparison of All Spinal Segments Kinematics ın Patients With Chronic Low Back Pain and Asymptomatic Individuals ın Three Planes During Activities of Daily Living
Brief Title: Assessment of All Spine Segments ın Individuals With Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sumeyye Zehra Guler, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HU-FTR-SZK-01
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: Rehabilitation; Kinematics; Activities of Daily Living
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Low back pain group and healthy group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Back Pain Group (Experimental): Low back pain group will be evaluated the kinematics of all spine segments in 3 planes while performing the tasks that patients with chronic low back pain often describe as painful in their daily lives,
  Interventions: Other: Low back pain group
- Healthy Group (Active Comparator): Healthy Group's results will be compared them with low back pain group
  Interventions: Other: Healthy group

INTERVENTIONS:
Other: Low back pain group — The low back pain group will be evaluated the kinematics of all spine segments in 3 planes while performing the tasks that patients with chronic low back pain often describe as painful in their daily lives such as walking, stepping up, standing up, bending and lifting. Using Inertial Measurement Sensors that provide valid and reliable will evaluate the kinematics of all spine
  Arms: Low Back Pain Group
Other: Healthy group — Low back pain kinematics compare them with asymptomatic kontrols
  Arms: Healthy Group

SUMMARY:
The aim of the study is to evaluate the kinematics of all spine segments in 3 planes and compare them with asymptomatic controls using wearable technology while performing functional tasks that patients with chronic low back pain often describe as painful in their daily lives.

DETAILED DESCRIPTION:
Low back pain is an important global health problem, with 84% of the population having at least one episode of low back pain in their lifetime and 23% developing a chronic form. It has been shown in many studies that the quality of life of individuals with low back pain is seriously reduced due to problems such as depression, anxiety, attention problems, sleep disorders, and social isolation. Low back pain has serious negative effects on national economies all over the world due to incapacity and increased medical expenses. According to the International Classification System of Health, individuals with low back pain often evaluated activities such as maintaining body position, changing basic body position, lifting objects, and walking as painful in their daily lives. Studies show that patients exhibit maladaptive spinal movement strategies that include increased trunk muscle activity and decreased trunk mobility to prevent further pain or injury during these activities. It was concluded that there was no difference in lordosis angles in people with low back pain compared to healthy controls, but there was a decrease in the lumbar range of motion in all directions of motion and they moved more slowly. It is seen that most of the studies focus only on the lumbar spine while evaluating functional activities, while other segments of the spine are ignored. The limited number of studies examining other segments concluded that the angle changes did not occur only in the lumbar spine and emphasized the importance of examining other segments together. For example, in a study conducted in individuals with low back pain and healthy individuals, it was found that during the task of step-up with three different step heights, patients exhibited more extension and less flexion in the upper thoracic joints in the sagittal plane, and it was recommended to examine the head movements in future studies. The same study also noted smaller lower thoracic and upper lumbar range of motion in patients in the frontal plane. According to these results, it can be said that examining functional activities in only one plane is insufficient due to the multifaceted nature of movement in individuals with low back pain. Defining spinal angles in different planes, examining different functional activities, and evaluating the spine as a whole are necessary to understand and effectively rehabilitate the changing spinal kinematics in low back pain. With the developing technology, many kinematic analysis methods have emerged to analyze the movement of body segments. Among these, Inertial Measurement Sensors have become effective tools for objective and quantitative evaluation due to their low cost, accuracy and portability. According to this information, in this study, it aim to evaluate the kinematics of all spine segments in 3 planes and compare them with asymptomatic controls while performing the tasks that patients with chronic low back pain often describe as painful in their daily lives, using these sensors that provide valid and reliable results for the kinematic analysis of functional activities. At the end of the study, it is expected that the motion patterns of the cervical, upper-lower thoracic, and upper-lower lumbar segments in 3 planes may differ kinematically in individuals with low back pain compared to healthy individuals, and the movement of the lumbar region in 3 planes may be affected by cervical and/or thoracic region movement. These results will guide the understanding of multifactorial low back pain and will enable the determination and implementation of appropriate preventive and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

For the low back pain group:

* Individuals aged 18-55 with non-specific chronic low back pain
* Individuals who have been experiencing pain for more than 3 months
* Individuals whose pain intensity is above 3 on the Visual Analog Scale

For the healthy group:

- Individuals aged 18-55 with no history of low back pain lasting more than 1 week for 6 months prior to the study

Exclusion Criteria:

* Current rheumatological or neurological diseases
* Recent or current pregnancy
* History of tumors or spine fractures
* Known spinal defects or surgery history
* Body mass index over 30 kg/m²

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the kinematics of the all spine during walking | two months
  Kinematic evaluations of functional activities will be performed using MVN Awinda (XSens Technologies B.V. Enschede, Netherlands) Inertial measurement unit sensors for walking. Angular data in the atlanto-occipital, C7-T1, T8-T9, T12-L1, L3-L4, and L5-S1 segments will be recorded in 3-dimensional. Participants will walk on a 10-meter walking path.
Evaluation of the kinematics of the all spine during Bending Forward and Lifting Objects | two months
  Kinematic evaluations of functional activities will be performed using MVN Awinda (XSens Technologies B.V. Enschede, Netherlands) Inertial measurement unit sensors for Bending Forward and Lifting Objects. The box (5 kilograms ) will be centered 15 centimeter in front of the participants' toes. Spinal kinematics will be analyzed from bending forward to lift the box, to holding the box in front of the hips and standing straight.
Evaluation of the kinematics of the all spine during Standing from Sitting | two months
  Kinematic evaluations of functional activities will be performed using MVN Awinda (XSens Technologies B.V. Enschede, Netherlands) Inertial measurement unit sensors for Standing from Sitting. Participants will stand up with their arms crossed over their chest at their preferred pace.
Evaluation of the kinematics of the all spine during Climbing Step | two months
  Kinematic evaluations of functional activities will be performed using MVN Awinda (XSens Technologies B.V. Enschede, Netherlands) Inertial measurement unit sensors for Climbing Step. Each participant will be asked to step onto a single 24 centimeter tall rectangular step placed ~13 centimeter from the big toe at a self-selected pace

SECONDARY OUTCOMES:
Spine Normal Joint Movement evaluation | two months
  Lumbar Spine Normal Joint Movement of Flexion, Extension, Lateral Flexion and Rotation movements will be evaluated by goniometric measurement.
Pain intensity: Visual Analog Scale | two months
  It is one of the pain rating scales. The pain Visual Analog Scale is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions.It is a straight horizontal line of fixed length, usually 100 milimeters. The ends are defined as the extreme limits of the parameter to be measured(pain) oriented from the left (worst) to the right (best).
Oswestry Disability Index | two months
  It is an important tool that researchers use to measure a patient's permanent functional disability. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. The higher scores indicate an increasing degree of disability.
Fear of movement: Tampa Kinesiophobia Scale | two months
  It is a self-reported questionnaire that quantifies fear of movement, or (re)injury. Individual item scores range from 1-4, with the negatively worded items (4,8,12,16) having a reverse scoring (4-1). The 17 item Tampa total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Zehra Güler, MSc, Principal Investigator — +90 5079320390
Locations (1):
- Hacettepe university, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell K, Porter M, Anderson L, Phillips C, Arceo G, Montz B, Levy S, Gombatto SP. Differences in lumbar spine and lower extremity kinematics in people with and without low back pain during a step-up task: a cross-sectional study. BMC Musculoskelet Disord. 2017 Aug 25;18(1):369. doi: 10.1186/s12891-017-1721-z. PMID 28841866
- [Background] Gombatto SP, Brock T, DeLork A, Jones G, Madden E, Rinere C. Lumbar spine kinematics during walking in people with and people without low back pain. Gait Posture. 2015 Oct;42(4):539-44. doi: 10.1016/j.gaitpost.2015.08.010. Epub 2015 Sep 3. PMID 26380913
- [Background] Papi E, Bull AMJ, McGregor AH. Spinal segments do not move together predictably during daily activities. Gait Posture. 2019 Jan;67:277-283. doi: 10.1016/j.gaitpost.2018.10.031. Epub 2018 Oct 29. PMID 30391750
- [Background] Laird RA, Keating JL, Ussing K, Li P, Kent P. Does movement matter in people with back pain? Investigating 'atypical' lumbo-pelvic kinematics in people with and without back pain using wireless movement sensors. BMC Musculoskelet Disord. 2019 Jan 18;20(1):28. doi: 10.1186/s12891-018-2387-x. PMID 30658610
- [Background] Saito H, Watanabe Y, Kutsuna T, Futohashi T, Kusumoto Y, Chiba H, Kubo M, Takasaki H. Spinal movement variability associated with low back pain: A scoping review. PLoS One. 2021 May 24;16(5):e0252141. doi: 10.1371/journal.pone.0252141. eCollection 2021. PMID 34029347
- [Background] Dogan M, Kocak M, Onursal Kilinc O, Ayvat F, Sutcu G, Ayvat E, Kilinc M, Unver O, Aksu Yildirim S. Functional range of motion in the upper extremity and trunk joints: Nine functional everyday tasks with inertial sensors. Gait Posture. 2019 May;70:141-147. doi: 10.1016/j.gaitpost.2019.02.024. Epub 2019 Feb 25. PMID 30875600
- [Background] Papi E, Bull AMJ, McGregor AH. Is there evidence to use kinematic/kinetic measures clinically in low back pain patients? A systematic review. Clin Biomech (Bristol). 2018 Jun;55:53-64. doi: 10.1016/j.clinbiomech.2018.04.006. Epub 2018 Apr 11. PMID 29684790
- [Background] Fong DT, Chan YY. The use of wearable inertial motion sensors in human lower limb biomechanics studies: a systematic review. Sensors (Basel). 2010;10(12):11556-65. doi: 10.3390/s101211556. Epub 2010 Dec 16. PMID 22163542
- [Background] Christe G, Redhead L, Legrand T, Jolles BM, Favre J. Multi-segment analysis of spinal kinematics during sit-to-stand in patients with chronic low back pain. J Biomech. 2016 Jul 5;49(10):2060-2067. doi: 10.1016/j.jbiomech.2016.05.015. Epub 2016 May 20. PMID 27262182
- [Background] Christe G, Aussems C, Jolles BM, Favre J. Patients With Chronic Low Back Pain Have an Individual Movement Signature: A Comparison of Angular Amplitude, Angular Velocity and Muscle Activity Across Multiple Functional Tasks. Front Bioeng Biotechnol. 2021 Nov 15;9:767974. doi: 10.3389/fbioe.2021.767974. eCollection 2021. PMID 34869281
- [Background] Christe G, Rochat V, Jolles BM, Favre J. Lumbar and thoracic kinematics during step-up: Comparison of three-dimensional angles between patients with chronic low back pain and asymptomatic individuals. J Orthop Res. 2020 Jun;38(6):1248-1256. doi: 10.1002/jor.24575. Epub 2020 Jan 7. PMID 31879969
- [Background] Aartun E, Axen I, Mior S, Roe Y, Hondras M, Kretz L, Cote P. Contextualizing the lived experiences of patients with low back pain from different countries according to the ICF framework. J Rehabil Med. 2021 May 11;53(5):jrm00189. doi: 10.2340/16501977-2819. PMID 33778896